CLINICAL TRIAL: NCT05987826
Title: Furmonertinib Mesylate Neoadjuvant Treatment of Resectable Stage Ⅱ-ⅢB Non-small Cell Lung Cancer Patients With Epidermal Growth Factor Receptor（EGFR）Sensitive Mutation：a Prospective，Muliticenter，Open Label，Phase Ⅱ Single-arm Study
Brief Title: Study of Furmonertinib as Neoadjuvant Therapy for Resectable Stage Ⅱ-ⅢB EGFR Sensitive Mutant NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Xuhui Central Hospital, Shanghai (Other); Shanghai Minhang Central Hospital (Other); Shanghai Zhongshan Hospital Qingpu Branch (Unknown); Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-170R
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: furmonertinib; neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (AST2818) 80mg QD group (Experimental): All patients enrolled into this study will receive furmonertinib 80mg for 8 weeks neoadjuvant therapy before surgery.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 80mg QD oral 8 weeks.
  Other Names: Furmonertinib(AST2818)

SUMMARY:
EGFR-TKI has firmly established itself as a first-line treatment for advanced lung cancer with EGFR-sensitive mutations, and the ADAURA study has added to its indications for use as postoperative adjuvant therapy in early- and mid-stage lung cancer.However, clinical data on neoadjuvant EGFR-TKI therapy are still incomplete. A phase II clinical study, CTONG1103, currently ongoing, comparing the efficacy of the first generational EGFR-TKI erlotinib and gemcitabine combined with cisplatin as neoadjuvant therapy for stage IIIA-N2 EGFR mutation-positive non-small-cell lung cancer, did not yield significantly positive objective remission rate (ORR) results.

Furmonertinib is a third-generation Epidermal Growth Factor Receptor (EGFR) tyrosine kinase inhibitor (TKI) that targets Epidermal Growth Factor Receptor (EGFR) mutations.Furmonertinib demonstrates definite efficacy and favorable safety in first-line EGFR-sensitive mutations and EGFR T790M Mutations in second-line and late-line treatment of advanced NSCLC.The aim of this study was to explore the efficacy and safety of furmonertinib neoadjuvant therapy for resectable stage II-IIIB EGFR-sensitive mutant non-small cell lung cancer efficacy and safety. Patinents are planned to be recruited from five centers in China. Eligible patients will receive furmonertinib neoadjuvant therapy for 8 weeks to evaluate the efficacy and safety of furmonnertinib neoadjuvant.

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

* 1）Provide informed consent prior to any study specific procedures
* 2）at least 18 years of age，not more than 75 years
* 3）Histology or cytology diagnose of non-small cell lung cancer within 60 days
* 4）ECOG PS of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks
* 5）Stage II-IIIB NSCLC that is expected to be resectable, as assessed by the investigator (8 thUICCTNM staging), with stage IIIB only including cT3N2M0 patients
* 6）According to RECIST 1.1, patients have at least one measureable tumor lesion (The longest axis ≥10mm)
* 7）EGFR mutation positive (exon 19 deletions or exon 21 L858R, with or without other EGFR mutations)
* 8）Without prior anti-tumor treatment
* 9) Withe adequate organ function of hematology, liver and kidney
* 10）Using adequate and effective contraception, Male patients should be use condoms; women should refrain from breastfeeding and have a negative pregnancy test prior to the first administration of the study drug if within during child-bearing age

Exclusion Criteria:

* 1）Dual or multiple primary NSCLC
* 2）Any prior anti-tumor treatment
* 3）With history of other malignancy except for radical resected tumors without recurrence for 5 years or more
* 4）History of interstitial lung disease or with relative risk factors
* 5）Diseases or clinical states with severe abnormalities of gastrointestinal function that may interfere with the ingestion, transit, or absorption of the study drug.e.g., inability to take medication orally, uncontrolled nausea and vomiting
* 6）Use of strong CYP3A4 inhibitors within 7 days or strong CYP3A4 inducers within 21 days before enrolment; use of traditional Chinese medicine with anti-tumor effect within 21 days before enrolment
* 7）With severe or uncontrolled systemic disease such as uncontrolled hypertention, diabetes mellitus, chronic heart failure, unstable angina, myocardial infarction within 1 year, active hemorrhage, active HBV/HCV/HIV or other infections requiring infusion treatment
* 8）Prolongation of ECG QTc or with relative risk factors
* 9）psychopath and/or mental illness
* 10）Pre-existing or coexisting bleeding disorders
* 11）Women with pregnancy or breastfeeding
* 12）Allergic to study drugs or any component
* 13）Other conditions that, in the opinion of the investigator, make participation in this trial inappropriate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | Approximately 8 weeks following the first dose of study drug
  According to RECIST 1.1 criteria, after 8 weeks of neoadjuvant therapy with furmonertinib CT scans scans assessed the proportion of patients in partial and complete remission.

SECONDARY OUTCOMES:
Main Pathological Response（MPR） | Approximately 12 weeks following the first dose of study drug
  Proportion of resected specimens with ≤10% residual tumor cells assessed by surgical specimen pathology
Pathological Complete Response Rate（pCR) | Approximately 12 weeks following the first dose of study drug
  The proportion of patients with pathological response rate in the resected tumor.
Pathological Nodal Downstaging Rate | Approximately 12 weeks following the first dose of study drug
  Neoadjuvant confirmed by pathologic evaluation of tumors and other tissues removed during surgery Percentage of patients downregulated from lymph node-positive to negative after treatment
Delayed Surgery Rate | Approximately 12 weeks following the first dose of study drug
  Proportion of surgeries performed 2 weeks after the last dose of furmonertinib because of adverse drug reactions and other reasons.
Rate of R0 Resection | Approximately 12 weeks following the first dose of study drug
  The proportion of patients with R0 resection.
Percentage of minimally invasive mid-rotation open chest | Approximately 12 weeks following the first dose of study drug
  Proportion of minimally invasive surgeries converted to open thoracic for various reasons
Incidence of adverse drug events (AE) | Approximately 12 weeks following the first dose of study drug
  Unfavorable clinical events in the course of drug treatment

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Herbst RS, Heymach JV, Lippman SM. Lung cancer. N Engl J Med. 2008 Sep 25;359(13):1367-80. doi: 10.1056/NEJMra0802714. No abstract available. PMID 18815398
- [Background] Rami-Porta R, Asamura H, Travis WD, Rusch VW. Lung cancer - major changes in the American Joint Committee on Cancer eighth edition cancer staging manual. CA Cancer J Clin. 2017 Mar;67(2):138-155. doi: 10.3322/caac.21390. Epub 2017 Jan 31. PMID 28140453
- [Background] Goldstraw P, Chansky K, Crowley J, Rami-Porta R, Asamura H, Eberhardt WE, Nicholson AG, Groome P, Mitchell A, Bolejack V; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for Revision of the TNM Stage Groupings in the Forthcoming (Eighth) Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Jan;11(1):39-51. doi: 10.1016/j.jtho.2015.09.009. PMID 26762738
- [Background] Coate LE, John T, Tsao MS, Shepherd FA. Molecular predictive and prognostic markers in non-small-cell lung cancer. Lancet Oncol. 2009 Oct;10(10):1001-10. doi: 10.1016/S1470-2045(09)70155-X. PMID 19796752
- [Background] Pignon JP, Tribodet H, Scagliotti GV, Douillard JY, Shepherd FA, Stephens RJ, Dunant A, Torri V, Rosell R, Seymour L, Spiro SG, Rolland E, Fossati R, Aubert D, Ding K, Waller D, Le Chevalier T; LACE Collaborative Group. Lung adjuvant cisplatin evaluation: a pooled analysis by the LACE Collaborative Group. J Clin Oncol. 2008 Jul 20;26(21):3552-9. doi: 10.1200/JCO.2007.13.9030. Epub 2008 May 27. PMID 18506026
- [Background] NSCLC Meta-analysis Collaborative Group. Preoperative chemotherapy for non-small-cell lung cancer: a systematic review and meta-analysis of individual participant data. Lancet. 2014 May 3;383(9928):1561-71. doi: 10.1016/S0140-6736(13)62159-5. Epub 2014 Feb 25. PMID 24576776
- [Background] Cancer Genome Atlas Research Network. Comprehensive genomic characterization of squamous cell lung cancers. Nature. 2012 Sep 27;489(7417):519-25. doi: 10.1038/nature11404. Epub 2012 Sep 9. PMID 22960745
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular profiling of lung adenocarcinoma. Nature. 2014 Jul 31;511(7511):543-50. doi: 10.1038/nature13385. Epub 2014 Jul 9. PMID 25079552
- [Background] George J, Lim JS, Jang SJ, Cun Y, Ozretic L, Kong G, Leenders F, Lu X, Fernandez-Cuesta L, Bosco G, Muller C, Dahmen I, Jahchan NS, Park KS, Yang D, Karnezis AN, Vaka D, Torres A, Wang MS, Korbel JO, Menon R, Chun SM, Kim D, Wilkerson M, Hayes N, Engelmann D, Putzer B, Bos M, Michels S, Vlasic I, Seidel D, Pinther B, Schaub P, Becker C, Altmuller J, Yokota J, Kohno T, Iwakawa R, Tsuta K, Noguchi M, Muley T, Hoffmann H, Schnabel PA, Petersen I, Chen Y, Soltermann A, Tischler V, Choi CM, Kim YH, Massion PP, Zou Y, Jovanovic D, Kontic M, Wright GM, Russell PA, Solomon B, Koch I, Lindner M, Muscarella LA, la Torre A, Field JK, Jakopovic M, Knezevic J, Castanos-Velez E, Roz L, Pastorino U, Brustugun OT, Lund-Iversen M, Thunnissen E, Kohler J, Schuler M, Botling J, Sandelin M, Sanchez-Cespedes M, Salvesen HB, Achter V, Lang U, Bogus M, Schneider PM, Zander T, Ansen S, Hallek M, Wolf J, Vingron M, Yatabe Y, Travis WD, Nurnberg P, Reinhardt C, Perner S, Heukamp L, Buttner R, Haas SA, Brambilla E, Peifer M, Sage J, Thomas RK. Comprehensive genomic profiles of small cell lung cancer. Nature. 2015 Aug 6;524(7563):47-53. doi: 10.1038/nature14664. Epub 2015 Jul 13. PMID 26168399
- [Background] Weinstein IB. Cancer. Addiction to oncogenes--the Achilles heal of cancer. Science. 2002 Jul 5;297(5578):63-4. doi: 10.1126/science.1073096. No abstract available. PMID 12098689
- [Background] Fernandez-Cuesta L, Plenker D, Osada H, Sun R, Menon R, Leenders F, Ortiz-Cuaran S, Peifer M, Bos M, Dassler J, Malchers F, Schottle J, Vogel W, Dahmen I, Koker M, Ullrich RT, Wright GM, Russell PA, Wainer Z, Solomon B, Brambilla E, Nagy-Mignotte H, Moro-Sibilot D, Brambilla CG, Lantuejoul S, Altmuller J, Becker C, Nurnberg P, Heuckmann JM, Stoelben E, Petersen I, Clement JH, Sanger J, Muscarella LA, la Torre A, Fazio VM, Lahortiga I, Perera T, Ogata S, Parade M, Brehmer D, Vingron M, Heukamp LC, Buettner R, Zander T, Wolf J, Perner S, Ansen S, Haas SA, Yatabe Y, Thomas RK. CD74-NRG1 fusions in lung adenocarcinoma. Cancer Discov. 2014 Apr;4(4):415-22. doi: 10.1158/2159-8290.CD-13-0633. Epub 2014 Jan 27. PMID 24469108
- [Background] Nakaoku T, Tsuta K, Ichikawa H, Shiraishi K, Sakamoto H, Enari M, Furuta K, Shimada Y, Ogiwara H, Watanabe S, Nokihara H, Yasuda K, Hiramoto M, Nammo T, Ishigame T, Schetter AJ, Okayama H, Harris CC, Kim YH, Mishima M, Yokota J, Yoshida T, Kohno T. Druggable oncogene fusions in invasive mucinous lung adenocarcinoma. Clin Cancer Res. 2014 Jun 15;20(12):3087-93. doi: 10.1158/1078-0432.CCR-14-0107. Epub 2014 Apr 11. PMID 24727320
- [Background] Kim Y, Hammerman PS, Kim J, Yoon JA, Lee Y, Sun JM, Wilkerson MD, Pedamallu CS, Cibulskis K, Yoo YK, Lawrence MS, Stojanov P, Carter SL, McKenna A, Stewart C, Sivachenko AY, Oh IJ, Kim HK, Choi YS, Kim K, Shim YM, Kim KS, Song SY, Na KJ, Choi YL, Hayes DN, Kim J, Cho S, Kim YC, Ahn JS, Ahn MJ, Getz G, Meyerson M, Park K. Integrative and comparative genomic analysis of lung squamous cell carcinomas in East Asian patients. J Clin Oncol. 2014 Jan 10;32(2):121-8. doi: 10.1200/JCO.2013.50.8556. Epub 2013 Dec 9. PMID 24323028
- [Background] Yarden Y, Sliwkowski MX. Untangling the ErbB signalling network. Nat Rev Mol Cell Biol. 2001 Feb;2(2):127-37. doi: 10.1038/35052073. PMID 11252954
- [Background] De Luca A, Carotenuto A, Rachiglio A, Gallo M, Maiello MR, Aldinucci D, Pinto A, Normanno N. The role of the EGFR signaling in tumor microenvironment. J Cell Physiol. 2008 Mar;214(3):559-67. doi: 10.1002/jcp.21260. PMID 17894407
- [Background] Jimeno A, Hidalgo M. Pharmacogenomics of epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors. Biochim Biophys Acta. 2006 Dec;1766(2):217-29. doi: 10.1016/j.bbcan.2006.08.008. Epub 2006 Sep 12. PMID 17045403
- [Background] Mosesson Y, Yarden Y. Oncogenic growth factor receptors: implications for signal transduction therapy. Semin Cancer Biol. 2004 Aug;14(4):262-70. doi: 10.1016/j.semcancer.2004.04.005. PMID 15219619
- [Background] Ciardiello F, Tortora G. EGFR antagonists in cancer treatment. N Engl J Med. 2008 Mar 13;358(11):1160-74. doi: 10.1056/NEJMra0707704. No abstract available. PMID 18337605
- [Background] Woodburn JR. The epidermal growth factor receptor and its inhibition in cancer therapy. Pharmacol Ther. 1999 May-Jun;82(2-3):241-50. doi: 10.1016/s0163-7258(98)00045-x. PMID 10454201
- [Background] Hazan RB, Norton L. The epidermal growth factor receptor modulates the interaction of E-cadherin with the actin cytoskeleton. J Biol Chem. 1998 Apr 10;273(15):9078-84. doi: 10.1074/jbc.273.15.9078. PMID 9535896
- [Background] Ellerbroek SM, Halbleib JM, Benavidez M, Warmka JK, Wattenberg EV, Stack MS, Hudson LG. Phosphatidylinositol 3-kinase activity in epidermal growth factor-stimulated matrix metalloproteinase-9 production and cell surface association. Cancer Res. 2001 Mar 1;61(5):1855-61. PMID 11280738
- [Background] Lee SY, Kim MJ, Jin G, Yoo SS, Park JY, Choi JE, Jeon HS, Cho S, Lee EB, Cha SI, Park TI, Kim CH, Jung TH, Park JY. Somatic mutations in epidermal growth factor receptor signaling pathway genes in non-small cell lung cancers. J Thorac Oncol. 2010 Nov;5(11):1734-40. doi: 10.1097/JTO.0b013e3181f0beca. PMID 20881644
- [Background] Yun CH, Boggon TJ, Li Y, Woo MS, Greulich H, Meyerson M, Eck MJ. Structures of lung cancer-derived EGFR mutants and inhibitor complexes: mechanism of activation and insights into differential inhibitor sensitivity. Cancer Cell. 2007 Mar;11(3):217-27. doi: 10.1016/j.ccr.2006.12.017. PMID 17349580
- [Background] Kumar A, Petri ET, Halmos B, Boggon TJ. Structure and clinical relevance of the epidermal growth factor receptor in human cancer. J Clin Oncol. 2008 Apr 1;26(10):1742-51. doi: 10.1200/JCO.2007.12.1178. PMID 18375904
- [Background] Yang JC, Camidge DR, Yang CT, Zhou J, Guo R, Chiu CH, Chang GC, Shiah HS, Chen Y, Wang CC, Berz D, Su WC, Yang N, Wang Z, Fang J, Chen J, Nikolinakos P, Lu Y, Pan H, Maniam A, Bazhenova L, Shirai K, Jahanzeb M, Willis M, Masood N, Chowhan N, Hsia TC, Jian H, Lu S. Safety, Efficacy, and Pharmacokinetics of Almonertinib (HS-10296) in Pretreated Patients With EGFR-Mutated Advanced NSCLC: A Multicenter, Open-label, Phase 1 Trial. J Thorac Oncol. 2020 Dec;15(12):1907-1918. doi: 10.1016/j.jtho.2020.09.001. Epub 2020 Sep 9. PMID 32916310
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Final overall survival results from a randomised, phase III study of erlotinib versus chemotherapy as first-line treatment of EGFR mutation-positive advanced non-small-cell lung cancer (OPTIMAL, CTONG-0802). Ann Oncol. 2015 Sep;26(9):1877-1883. doi: 10.1093/annonc/mdv276. Epub 2015 Jul 3. PMID 26141208
- [Background] Cross DA, Ashton SE, Ghiorghiu S, Eberlein C, Nebhan CA, Spitzler PJ, Orme JP, Finlay MR, Ward RA, Mellor MJ, Hughes G, Rahi A, Jacobs VN, Red Brewer M, Ichihara E, Sun J, Jin H, Ballard P, Al-Kadhimi K, Rowlinson R, Klinowska T, Richmond GH, Cantarini M, Kim DW, Ranson MR, Pao W. AZD9291, an irreversible EGFR TKI, overcomes T790M-mediated resistance to EGFR inhibitors in lung cancer. Cancer Discov. 2014 Sep;4(9):1046-61. doi: 10.1158/2159-8290.CD-14-0337. Epub 2014 Jun 3. PMID 24893891
- [Background] Wu YL, Ahn MJ, Garassino MC, Han JY, Katakami N, Kim HR, Hodge R, Kaur P, Brown AP, Ghiorghiu D, Papadimitrakopoulou VA, Mok TSK. CNS Efficacy of Osimertinib in Patients With T790M-Positive Advanced Non-Small-Cell Lung Cancer: Data From a Randomized Phase III Trial (AURA3). J Clin Oncol. 2018 Sep 10;36(26):2702-2709. doi: 10.1200/JCO.2018.77.9363. Epub 2018 Jul 30. PMID 30059262
- [Background] Goss G, Tsai CM, Shepherd FA, Bazhenova L, Lee JS, Chang GC, Crino L, Satouchi M, Chu Q, Hida T, Han JY, Juan O, Dunphy F, Nishio M, Kang JH, Majem M, Mann H, Cantarini M, Ghiorghiu S, Mitsudomi T. Osimertinib for pretreated EGFR Thr790Met-positive advanced non-small-cell lung cancer (AURA2): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1643-1652. doi: 10.1016/S1470-2045(16)30508-3. Epub 2016 Oct 14. PMID 27751847
- [Background] Yang JC, Ahn MJ, Kim DW, Ramalingam SS, Sequist LV, Su WC, Kim SW, Kim JH, Planchard D, Felip E, Blackhall F, Haggstrom D, Yoh K, Novello S, Gold K, Hirashima T, Lin CC, Mann H, Cantarini M, Ghiorghiu S, Janne PA. Osimertinib in Pretreated T790M-Positive Advanced Non-Small-Cell Lung Cancer: AURA Study Phase II Extension Component. J Clin Oncol. 2017 Apr 20;35(12):1288-1296. doi: 10.1200/JCO.2016.70.3223. Epub 2017 Feb 21. PMID 28221867
- [Background] Ramalingam SS, Vansteenkiste J, Planchard D, Cho BC, Gray JE, Ohe Y, Zhou C, Reungwetwattana T, Cheng Y, Chewaskulyong B, Shah R, Cobo M, Lee KH, Cheema P, Tiseo M, John T, Lin MC, Imamura F, Kurata T, Todd A, Hodge R, Saggese M, Rukazenkov Y, Soria JC; FLAURA Investigators. Overall Survival with Osimertinib in Untreated, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2020 Jan 2;382(1):41-50. doi: 10.1056/NEJMoa1913662. Epub 2019 Nov 21. PMID 31751012
- [Background] Zhong WZ, Wang Q, Mao WM, Xu ST, Wu L, Shen Y, Liu YY, Chen C, Cheng Y, Xu L, Wang J, Fei K, Li XF, Li J, Huang C, Liu ZD, Xu S, Chen KN, Xu SD, Liu LX, Yu P, Wang BH, Ma HT, Yan HH, Yang XN, Zhou Q, Wu YL; ADJUVANT investigators. Gefitinib versus vinorelbine plus cisplatin as adjuvant treatment for stage II-IIIA (N1-N2) EGFR-mutant NSCLC (ADJUVANT/CTONG1104): a randomised, open-label, phase 3 study. Lancet Oncol. 2018 Jan;19(1):139-148. doi: 10.1016/S1470-2045(17)30729-5. Epub 2017 Nov 21. PMID 29174310
- [Background] Li N, Ou W, Ye X, Sun HB, Zhang L, Fang Q, Zhang SL, Wang BX, Wang SY. Pemetrexed-carboplatin adjuvant chemotherapy with or without gefitinib in resected stage IIIA-N2 non-small cell lung cancer harbouring EGFR mutations: a randomized, phase II study. Ann Surg Oncol. 2014 Jun;21(6):2091-6. doi: 10.1245/s10434-014-3586-9. Epub 2014 Mar 1. PMID 24585406
- [Background] Kappers I, Klomp HM, Burgers JA, Van Zandwijk N, Haas RL, van Pel R. Neoadjuvant (induction) erlotinib response in stage IIIA non-small-cell lung cancer. J Clin Oncol. 2008 Sep 1;26(25):4205-7. doi: 10.1200/JCO.2008.16.3709. No abstract available. PMID 18757336
- [Background] Wang Q, Wang H, Li P, Zhu H, He C, Wei B, Ma J, Ma Z. Erlotinib-based perioperative adjuvant therapy for a case of unresectable stage IIIA (N2) nonsmall cell lung cancer. Am J Med Sci. 2010 Oct;340(4):321-5. doi: 10.1097/MAJ.0b013e3181e59ac2. PMID 20601859
- [Background] Zhong WZ, Chen KN, Chen C, Gu CD, Wang J, Yang XN, Mao WM, Wang Q, Qiao GB, Cheng Y, Xu L, Wang CL, Chen MW, Kang X, Yan W, Yan HH, Liao RQ, Yang JJ, Zhang XC, Zhou Q, Wu YL. Erlotinib Versus Gemcitabine Plus Cisplatin as Neoadjuvant Treatment of Stage IIIA-N2 EGFR-Mutant Non-Small-Cell Lung Cancer (EMERGING-CTONG 1103): A Randomized Phase II Study. J Clin Oncol. 2019 Sep 1;37(25):2235-2245. doi: 10.1200/JCO.19.00075. Epub 2019 Jun 13. PMID 31194613
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Herbst RS, Sandler A. Bevacizumab and erlotinib: a promising new approach to the treatment of advanced NSCLC. Oncologist. 2008 Nov;13(11):1166-76. doi: 10.1634/theoncologist.2008-0108. Epub 2008 Nov 8. PMID 18997180
- [Background] Zhou Q, Xu CR, Cheng Y, Liu YP, Chen GY, Cui JW, Yang N, Song Y, Li XL, Lu S, Zhou JY, Ma ZY, Yu SY, Huang C, Shu YQ, Wang Z, Yang JJ, Tu HY, Zhong WZ, Wu YL. Bevacizumab plus erlotinib in Chinese patients with untreated, EGFR-mutated, advanced NSCLC (ARTEMIS-CTONG1509): A multicenter phase 3 study. Cancer Cell. 2021 Sep 13;39(9):1279-1291.e3. doi: 10.1016/j.ccell.2021.07.005. Epub 2021 Aug 12. PMID 34388377
- [Background] Li K, Cao X, Ai B, Xiao H, Huang Q, Zhang Z, Chu Q, Zhang L, Dai X, Liao Y. Salvage surgery following downstaging of advanced non-small cell lung cancer by targeted therapy. Thorac Cancer. 2021 Aug;12(15):2161-2169. doi: 10.1111/1759-7714.14044. Epub 2021 Jun 15. PMID 34128318
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] Deng H, Liu J, Cai X, Chen J, Rocco G, Petersen RH, Brunelli A, Ng CSH, D'Amico TA, Liang W, He J. Radical Minimally Invasive Surgery After Immuno-chemotherapy in Initially-unresectable Stage IIIB Non-small cell Lung Cancer. Ann Surg. 2022 Mar 1;275(3):e600-e602. doi: 10.1097/SLA.0000000000005233. PMID 34596079
- See also: Related Info — https://seer.cancer.gov/